CLINICAL TRIAL: NCT01491659
Title: A Randomised, Double-blind, Placebo-controlled Study to Evaluate the Effect and Safety of Idoform Plus on Bowel Side Effects in Healthy Subjects Treated With Amoxicillin/ Clavulanate
Brief Title: A Study to Evaluate the Effect and Safety of Idoform Plus on Bowel Side Effects in Healthy Subjects Treated With Amoxicillin/ Clavulanate
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Danisco/Dupont (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B4141002
Record Dates: First submitted 2011-12-05; First posted 2011-12-14 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Diarrhoea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin/clavulanate/Idoform Plus (Active Comparator)
  Interventions: Dietary Supplement: Idoform Plus
- Amoxicillin/clavulanate/Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Idoform Plus — orally once daily
  Arms: Amoxicillin/clavulanate/Idoform Plus
Dietary Supplement: Placebo — orally once daily
  Arms: Amoxicillin/clavulanate/Placebo

SUMMARY:
It is hypothesized that Idoform plus will recuce the occurence of gastrointestinal side effects related to the use of antibiotics

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers 18-70 years of age
* Subjects with normal gastrointestinal function
* Subjects willing to provide written informed consent

Exclusion Criteria:

* Subjects receiving antibiotic treatment within three months prior to inclusion in the study
* Pregnancy or planned pregnancy
* Breast feeding
* Subjects who are allergic to beta-lactam antibiotics, amoxicillin / clavulanate or its components
* Subjects with known renal insufficiency
* Subjects using products containing probiotics, fibers and/or prebiotics
* Subjects using proton pump inhibitors
* Subjects using H2 antagonists
* Subjects using antacids frequently

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Occurence of Antibiotic Associated Diarrhea | 17 days

SECONDARY OUTCOMES:
Duration of Antibiotic Associated Diarrhoea | 17 days
Occurrence of Antibiotic Associated Loose Stools (Types 5,6 or 7 on the Bristol Stool Chart) at Least Once During a Day | 17 days
Presence of Gastrointestinal Symptoms (Abdominal Pain; Bloating/Distension; Nausea/Upset Stomach), and the Severity of Each Symptom | 17 days
Changes in the Gut Microbiota Composition | 17 days
Changes in Markers of Antibiotic Resistance | 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4141002&StudyName=A%20Study%20to%20Evaluate%20the%20Effect%20and%20Safety%20of%20Idoform%20Plus%20on%20Bowel%20Side%20Effects%20in%20Healthy%20Subjects%20Treated%20With%20Amoxicillin/%20Clavul